CLINICAL TRIAL: NCT02230553
Title: Phase I/II Study With Lapatinib Plus Trametinib in Patients With Metastatic KRAS Mutant Non-small Cell Lung Cancer
Brief Title: Lapatinib Plus Trametinib in KRAS Mutant NSCLC
Acronym: M14LTK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL49551.031.14
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lapatinib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lapatinib + trametinib (Experimental): lapatinib: oral tablets, once daily trametinib: oral tablets, once daily
  Interventions: Drug: Lapatinib; Drug: trametinib

INTERVENTIONS:
Drug: Lapatinib
Drug: trametinib

SUMMARY:
This is an open-label phase I/II multi-center study consisting of two parts. Part A of this study is designed to identify the recommended phase 2 dose (RP2D) of lapatinib combined with trametinib in patients with metastatic KRASm and PIK3CA wild-type (PIK3CAwt) non-small cell lung cancer (NSCLC). Part B is designed to perform a randomized comparison of the lapatinib-trametinib combination versus standard of care therapy in patients with metastatic KRASm/PIK3CAwt NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of metastatic NSCLC; for PART B: treated with first line therapy for metastatic disease only.
* Written documentation of a known pathogenic KRAS (exon 2, 3 or 4) mutation and PIK3CA wild-type (exon 9 and 20)
* Age ≥ 18 years
* Able and willing to give written informed consent
* WHO performance status of 0 or 1 (part A and B)

Exclusion Criteria:

* Any treatment with investigational drugs within 30 days prior to receiving the first dose of investigational treatment.
* History of another primary malignancy
* Symptomatic or untreated leptomeningeal disease
* Symptomatic brain metastasis
* History of interstitial lung disease or pneumonitis
* Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients
* Retinal degenerative disease (hereditary retinal degeneration or age-related macular degeneration), or a history of uveitis, retinal vein occlusion, central serous retinopathy, or retinal detachment
* Patients with left ventricular ejection fraction (LVEF) < 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose-limiting toxicities | 1.5 years
progression free survival | 2.5 years
overall response rate | 2.5 years

SECONDARY OUTCOMES:
Incidence and severity of adveres events | 2.5 years
Plasma concentration | 2.5 years
Duration of response | 2.5 years
Time to response | 2.5 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: F Opdam, MD, PhD, Study Director — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands